CLINICAL TRIAL: NCT04677660
Title: A Phase 1/2, Randomized, Observer-Blind, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of TAK-919 by Intramuscular Injection in Healthy Japanese Male and Female Adults Aged 20 Years and Older (COVID-19)
Brief Title: A Study of TAK-919 in Healthy Japanese Adults (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAK-919-1501; U1111-1261-9040 (Other: WHO); jRCT2071200069 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-12-18; First posted 2020-12-21 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-02

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAK-919 (Experimental): TAK-919 0.5 mL, intramuscular injection in the upper arm
  Interventions: Biological: TAK-919
- Placebo (Placebo Comparator): TAK-919 Matching Placebo, intramuscular injection in the upper arm
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TAK-919 — TAK-919 intramuscular injection
  Arms: TAK-919
Biological: Placebo — Placebo intramuscular injection
  Arms: Placebo

SUMMARY:
TAK-919 is a vaccine in development to protect people against Covid-19. The main aims of the study are to learn if TAK-919 can protect people from Covid-19 and to check for side effects from TAK-919.

At the first visit, the study doctor will check if each person can take part. Those who can take part will be chosen for 1 of 2 treatments by chance. Participants will either receive an injection of TAK-919 or a placebo in their arm. In this study, a placebo will look like the TAK-919 vaccine but will not have any medicine in it. 3 times as many participants will receive TAK-919 than placebo. Participants will receive 2 injections of TAK-919 or placebo, 28 days apart.

Participants will be asked to record their temperature and any medical problems in an electronic diary for up to 7 days after each injection.

During the study, participants will visit the clinic for regular check-ups, blood tests, and sometimes for nose swab samples. When all participants have visited their clinic 28 days after their 2nd injection, the study sponsor (Takeda) will check how many participants have made enough antibodies to protect them against Covid-19.

The participants will stay in the study for up to 12 months after they have had their 2nd injection. During this time, the study doctors will continue to check how many participants have made enough antibodies to protect them against Covid-19. Also, they will check if participants have any more side effects from TAK-919 or the placebo.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-919. TAK-919 is being tested to prevent infectious disease caused by Severe Acute Respiratory Syndrome coronavirus-2 (SARS-CoV-2). This study will look at the safety and immunogenicity of 2 doses of TAK-919 by intramuscular (IM) injection in healthy Japanese male and female adults, given 28 days apart.

The study will enroll approximately 200 healthy volunteers. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-919 0.5 mL
* Placebo- this is an injection that looks like the study drug but has no active ingredient

All participants will be asked to take intramuscular injection in the upper arm twice throughout the study.

This multi-center trial will be conducted in Japan. The overall time to participate in this study is 12 months from the second vaccination. Participants will make multiple visits to the clinic and will be contacted by telephone or a final visit after the last vaccination for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese male and female participants.
2. Participants who understand and are willing to comply with trial procedures and are available for the duration of follow up.

Exclusion Criteria:

1. Participants who received any other SARS-CoV-2 or other experimental novel coronavirus vaccine prior to the trial.
2. Participants who have close contact of anyone known to have COVID-19 within 30 days prior to vaccine administration.
3. Participants who were tested positive for SARS-CoV-2 prior to the trial or on the test before the vaccination.
4. Participants who are on current treatment with other investigational agents for prophylaxis of COVID 19.
5. Participants who traveled outside of Japan in the 30 days prior to the trial participation.
6. Participants with a clinically significant active infection (as assessed by the Investigator) or oral temperature >= 38 degree Celsius within 3 days of the vaccination.
7. Participants with a known hypersensitivity or allergy to any of the IMP components.
8. Participants with any illness or history of any illness that, in the opinion of the Investigator, might interfere with the results of the trial or pose additional risk to the participants due to participation in the trial.
9. Participants with known or suspected impairment/alteration of immune function, including history of any autoimmune disease or neuro-inflammatory disease.
10. Abnormalities of splenic or thymic function.
11. Participants with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
12. Participants with any serious chronic or progressive disease (eg, neoplasm, insulin dependent diabetes, cardiac, renal, or hepatic disease).
13. Participants with BMI >= 30 kg/m^2 (BMI=weight in kg/height in meters^2).
14. Participants participating in any clinical trial with another investigational product within 30 days prior to the vaccination or intend to participate in another clinical trial at any time during the conduct of this trial.
15. Participants who received or plan to receive any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to trial dose administration.
16. Participants with acute or chronic clinically significant disease including pulmonary, cardiovascular, hepatic, or renal abnormality evaluated by physical examination.
17. Participants involved in the trial conduct or their first-degree relatives.
18. Participants who are with or have history of hepatitis B and hepatitis C infection, or with known human immunodeficiency virus (HIV) infection or HIV-related disease..
19. Female participants who are pregnant or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Sumida Hospital, Sumida-ku, Tokyo
  - PS Clinic, Fukuoka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Masuda T, Murakami K, Sugiura K, Sakui S, Philip Schuring R, Mori M. A phase 1/2 randomised placebo-controlled study of the COVID-19 vaccine mRNA-1273 in healthy Japanese adults: An interim report. Vaccine. 2022 Mar 18;40(13):2044-2052. doi: 10.1016/j.vaccine.2022.02.030. Epub 2022 Feb 8. PMID 35177302
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5ff2d498565ce300294c6ab5

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan from 07 January 2021 to 22 February 2022.
Pre-assignment Details: Healthy Japanese participants were enrolled to receive two doses of TAK-919 or saline placebo by intramuscular injection on Day 1 (first vaccination) and Day 29 (second vaccination).
Groups:
- Placebo: TAK-919 placebo-matching, injection, intramuscularly, once on Days 1 and 29 in healthy participants.
- TAK-919 0.5 mL: TAK-919 0.5 milliliter (mL), injection, intramuscularly, once on Days 1 and 29 in healthy participants.
Period: Overall Study
Arm/Group | Placebo | TAK-919 0.5 mL
Started | 50 | 150
Completed | 7 | 137
Not Completed | 43 | 13
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Chose Publicly Available Vaccine | 43 | 10

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Groups:
- TAK-919 0.5 mL: TAK-919 0.5 mL, injection, intramuscularly, once on Days 1 and 29 in healthy participants.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-919 0.5 mL | Total
Number analyzed (Participants) | 50 | 150 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (14.18) | 53.3 (15.67) | 53.1 (15.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 65 | 88
  Male | 27 | 85 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 50 | 150 | 200
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 50 | 150 | 200
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 62.49 (10.870) | 61.05 (9.918) | 61.41 (10.156)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 163.09 (8.501) | 164.83 (8.549) | 164.39 (8.549)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 23.35 (2.595) | 22.39 (2.653) | 22.63 (2.665)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) for Six Subsequent Days Following First Vaccination
Description: Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for six subsequent days following first vaccination. Solicited local AEs included injection site pain, erythema/redness, swelling, induration, and axillary (underarm) swelling or tenderness ipsilateral to the side of injection.
Time Frame: Up to Day 7 (6 subsequent days after first vaccination on Day 1)
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants
  Injection Site Pain | 6.0 | 82.7
  Erythema/ Redness | 0.0 | 2.0
  Swelling | 0.0 | 10.7
  Induration | 0.0 | 6.0
  Lymphadenopathy (Axillary Swelling or Tenderness at Same Side of Injection Site) | 4.0 | 11.3

2. Primary Outcome: Percentage of Participants With Solicited Local AEs for Six Subsequent Days Following Second Vaccination
Description: Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for six subsequent days following second vaccination. Solicited local AEs included injection site pain, erythema/redness, swelling, induration, and axillary (underarm) swelling or tenderness ipsilateral to the side of injection.
Time Frame: Up to Day 35 (6 subsequent days after second vaccination on Day 29)
Population: The safety analysis set included all participants who received at least 1 dose of the treatment. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
percentage of participants
  Injection Site Pain | 2.0 | 85.0
  Erythema/ Redness | 0.0 | 17.7
  Swelling | 0.0 | 16.3
  Induration | 0.0 | 12.9
  Lymphadenopathy (Axillary Swelling or Tenderness at Same Side of Injection Site) | 6.0 | 10.2

3. Primary Outcome: Percentage of Participants With Solicited Systemic AEs for Six Subsequent Days Following First Vaccination
Description: Solicited systemic AEs were pre-defined AEs for which participants were specifically questioned and which were noted by participants in their diary for six subsequent days following first vaccination. Solicited systemic AEs included headache, fatigue, myalgia, arthralgia, nausea/ vomiting, chills, fever.
Time Frame: Up to Day 7 (6 subsequent days after first vaccination on Day 1)
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants
  Headache | 0.0 | 13.3
  Fatigue | 10.0 | 18.7
  Myalgia | 4.0 | 37.3
  Arthralgia | 0.0 | 8.0
  Nausea/ Vomiting | 0.0 | 0.7
  Chills | 2.0 | 5.3
  Fever | 2.0 | 2.0

4. Primary Outcome: Percentage of Participants With Solicited Systemic AEs for Six Subsequent Days Following Second Vaccination
Description: Solicited systemic AEs were pre-defined AEs for which participants were specifically questioned and which were noted by participants in their diary for six subsequent days following second vaccination. Solicited systemic AEs included headache, fatigue, myalgia, arthralgia, nausea/ vomiting, chills, fever.
Time Frame: Up to Day 35 (6 subsequent days after second vaccination on Day 29)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
percentage of participants
  Headache | 10.0 | 47.6
  Fatigue | 8.0 | 63.3
  Myalgia | 10.0 | 49.7
  Arthralgia | 0.0 | 32.0
  Nausea/ Vomiting | 0.0 | 4.1
  Chills | 0.0 | 50.3
  Fever | 0.0 | 40.1

5. Primary Outcome: Percentage of Participants With Unsolicited AEs for 28 Days Following First Vaccination
Description: Unsolicited AEs were all AEs that were not pre-defined for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to Day 29 (28 days after first vaccination on Day 1)
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 18.0 | 20.7

6. Primary Outcome: Percentage of Participants With Unsolicited AEs for 28 Days Following Second Vaccination
Description: as for outcome 5
Time Frame: Up to Day 57 (28 days after second vaccination on Day 29)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
percentage of participants | 14.0 | 19.0

7. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Until Day 57
Description: Only unsolicited SAEs data was planned to be collected and assessed for the assessment of this outcome measure (OM) and solicited SAE was out of the scope of the assessment. Unsolicited SAEs were those AEs that were not pre-defined for which the participant is not specifically questioned in the participant diary. Percentage of participants with unsolicited SAEs until Day 57 was reported in this outcome measure.
Time Frame: Day 1 up to Day 57
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

8. Primary Outcome: Percentage of Participants With Medically-Attended Adverse Events (MAAEs) Until Day 57
Description: MAAEs were defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria. Only unsolicited MAAEs data was planned to be collected and assessed for the assessment of this OM and solicited MAAEs was out of the scope of the assessment. Unsolicited MAAEs were those AEs that were not pre-defined for which the participant is not specifically questioned in the participant diary. Percentage of participants with unsolicited MAAEs until Day 57 was reported in this outcome measure.
Time Frame: Day 1 up to Day 57
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 2.0 | 5.3

9. Primary Outcome: Percentage of Participants With Any AE Leading to Discontinuation of Vaccination
Description: Only unsolicited AE leading to discontinuation of vaccination data was planned to be collected and assessed for the assessment of this OM and solicited AE leading to discontinuation of vaccination was out of the scope of the assessment. Unsolicited AEs were those AEs that were not pre-defined for which the participant is not specifically questioned in the participant diary. Percentage of participants with any unsolicited AE leading to discontinuation of vaccination was reported in this outcome measure.
Time Frame: Day 1 up to Day 57
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 1.3

10. Primary Outcome: Percentage of Participants With Any AE Leading to Participant's Withdrawal From the Trial Until Day 57
Description: Only unsolicited AE leading to participant's withdrawal data was planned to be collected and assessed for the assessment of this OM and solicited AE leading to participant's withdrawal was out of the scope of the assessment. Unsolicited AEs were those AEs that were not pre-defined for which the participant is not specifically questioned in the participant diary. Percentage of participants with any unsolicited AE leading to participant's withdrawal from the trial until Day 57 was reported in this outcome measure.
Time Frame: Day 1 up to Day 57
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

11. Primary Outcome: Percentage of Participants With Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Infection Until Day 57
Time Frame: Day 1 up to Day 57
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

12. Primary Outcome: Geometric Mean Titers (GMT) of Serum Binding Antibody (bAb) Against SARS-CoV-2 on Day 57
Description: GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average for each group. Titer values measured as below lower limit of quantification (LLOQ) were imputed to a value that is half of the LLOQ. Titer values measured as above upper limit of quantification (ULOQ) were imputed at the ULOQ value. LLOQ=1 and ULOQ= 2052. GMT of serum bAb against SARS-CoV-2 was measured by ligand-binding assay specific to the SARS-CoV-2 spike (S) protein.
Time Frame: At Day 57
Population: The per-protocol-set (PPS) included participants who received at least one dose of the treatment and who had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary unit per milliliter (AU/mL)
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
arbitrary unit per milliliter (AU/mL) | 0.60 [0.53 to 0.67] | 813.05 [759.31 to 870.60]

13. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Serum bAb Against SARS-CoV-2 on Day 57
Description: The GMFR was calculated as the ratio of the post-vaccination titer level to the baseline titer level. Where baseline was defined as the last measurement taken before the first dose of study intervention. GMFR of serum bAb against SARS-CoV-2 was measured by ligand-binding assay specific to the SARS-CoV-2 S protein.
Time Frame: At Day 57
Population: The PPS included participants who received at least one dose of the treatment and who had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
fold change | 0.90 [0.83 to 0.99] | 1009.25 [865.11 to 1177.40]

14. Primary Outcome: Seroconversion Rate (SCR) of Serum bAb Against SARS-CoV-2 on Day 57
Description: SCR was defined as percentage of participants with a change from below limit of detection (LOD) or LLOQ to equal to or above LOD or LLOQ, OR, greater than or equal to (>=) 4-fold rises from baseline. LLOQ= 1, ULOQ= 2052. Baseline was defined as the last measurement taken before the first dose of study intervention. SCR of serum bAb against SARS-CoV-2 was measured by ligand-binding assay specific to the SARS-CoV-2 S protein.
Time Frame: At Day 57
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
percentage of participants | 2.0 [0.1 to 10.6] | 100.0 [97.5 to 100.0]

15. Secondary Outcome: Percentage of Participants With SAE Throughout the Trial
Description: Only unsolicited SAEs data was planned to be collected and assessed for the assessment of this OM and solicited SAE was out of the scope of the assessment. Unsolicited SAEs were those AEs that were not pre-defined for which the participant is not specifically questioned in the participant diary. Percentage of participants with unsolicited SAEs throughout the trial was reported in this outcome measure.
Time Frame: Day 1 up to Day 394
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

16. Secondary Outcome: Percentage of Participants With MAAEs Throughout the Trial
Description: MAAEs were defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria. Only unsolicited MAAEs data was planned to be collected and assessed for the assessment of this OM and solicited MAAEs was out of the scope of the assessment. Unsolicited MAAEs were those AEs that were not pre-defined for which the participant is not specifically questioned in the participant diary. Percentage of participants with unsolicited MAAEs throughout the trial was reported in this outcome measure.
Time Frame: Day 1 up to Day 394
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 4.0 | 14.7

17. Secondary Outcome: Percentage of Participants With Any AE Leading to Participant's Withdrawal From the Trial From the Day of Vaccination Throughout the Trial
Description: Only unsolicited AE leading to participant's withdrawal data was planned to be collected and assessed for the assessment of this OM and solicited AE leading to participant's withdrawal was out of the scope of the assessment. Unsolicited AEs were those AEs that were not pre-defined for which the participant is not specifically questioned in the participant diary. Percentage of participants with any unsolicited AE leading to participant's withdrawal from the trial from the day of vaccination throughout the trial was reported in this outcome measure.
Time Frame: Day 1 up to Day 394
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

18. Secondary Outcome: Percentage of Participants With SARS-CoV-2 Infection Throughout the Trial
Time Frame: Day 1 up to Day 394
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 1.3

19. Secondary Outcome: GMT of Serum bAb Against SARS-CoV-2 on Days 29, 43, 209 and 394
Description: GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average for each group. Titer values measured as below LLOQ were imputed to a value that is half of the LLOQ. Titer values measured as above ULOQ were imputed at the ULOQ value. LLOQ=1 and ULOQ= 2052 until Day 43; LLOQ= 1 and ULOQ= 20520 from Day 209 and later. GMT of serum bAb against SARS-CoV-2 was measured by ligand-binding assay specific to the SARS-CoV-2 S protein.
Time Frame: At Days 29, 43, 209 and 394
Population: The PPS included participants who received at least one dose of the treatment and who had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment. Here, "number analyzed" signifies those participants who were evaluable for this outcome measure at given timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
AU/mL
  Day 29 | 0.65 [0.57 to 0.74] | 140.72 [124.84 to 158.62]
  Day 43 | 0.62 [0.55 to 0.70] | 1021.71 [940.66 to 1109.73]
  Day 209: number analyzed (Participants) | 12 | 145
  Day 209 | 0.70 [0.51 to 0.96] | 116.97 [106.26 to 128.76]
  Day 394: number analyzed (Participants) | 7 | 134
  Day 394 | 1.28 [0.38 to 4.33] | 53.36 [46.74 to 60.92]

20. Secondary Outcome: GMFR of Serum bAb Against SARS-CoV-2 on Days 29, 43, 209 and 394
Description: as for outcome 13
Time Frame: At Days 29, 43, 209 and 394
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
fold change
  Day 29 | 0.99 [0.90 to 1.08] | 174.67 [148.72 to 205.16]
  Day 43 | 0.93 [0.87 to 1.00] | 1268.26 [1073.44 to 1498.43]
  Day 209: number analyzed (Participants) | 12 | 145
  Day 209 | 1.00 [0.81 to 1.24] | 145.97 [124.69 to 170.89]
  Day 394: number analyzed (Participants) | 7 | 134
  Day 394 | 1.71 [0.44 to 6.63] | 65.01 [53.96 to 78.32]

21. Secondary Outcome: SCR of Serum bAb Against SARS-CoV-2 on Days 29, 43, 209 and 394
Description: SCR was defined as percentage of participants with a change from below LOD or LLOQ to equal to or above LOD or LLOQ, OR >=4-fold rises from baseline. LLOQ= 1 and ULOQ= 2052 until Day 43; LLOQ= 1 and ULOQ= 20520 from Day 209 and later. Baseline was defined as the last measurement taken before the first dose of study intervention. SCR of serum bAb against SARS-CoV-2 was measured by ligand-binding assay specific to the SARS-CoV-2 S protein.
Time Frame: At Days 29, 43, 209 and 394
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
percentage of participants
  Day 29 | 6.0 [1.3 to 16.5] | 100.0 [97.5 to 100.0]
  Day 43 | 2.0 [0.1 to 10.6] | 100.0 [97.5 to 100.0]
  Day 209: number analyzed (Participants) | 12 | 145
  Day 209 | 8.3 [0.2 to 38.5] | 99.3 [96.2 to 100.0]
  Day 394: number analyzed (Participants) | 7 | 134
  Day 394 | 28.6 [3.7 to 71.0] | 97.0 [92.5 to 99.2]

22. Secondary Outcome: GMT of Serum Neutralizing Antibody (nAb) Against SARS-CoV-2 on Days 29, 43, 57, 209, and 394
Description: GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average for each group. Titer values measured as below LLOQ were imputed to a value that is half of the LLOQ. Titer values measured as above ULOQ were imputed at the ULOQ value. LLOQ= 159.79 and ULOQ= 11173.11. GMT of serum nAb against SARS-CoV-2 was measured by assay specific to wild-type virus.
Time Frame: At Days 29, 43, 57, 209, and 394
Population: PPS included participants in the FAS and who had evaluable immunogenicity data and did not have significant protocol deviations which influence the immunogenicity assessment. Here, "number analyzed" signifies those participants who were evaluable for this outcome measure at given timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: microneutralization titers (MN50)
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
microneutralization titers (MN50)
  Day 29: number analyzed (Participants) | 50 | 139
  Day 29 | 79.9 [79.9 to 79.9] | 202.4 [170.5 to 240.2]
  Day 43: number analyzed (Participants) | 50 | 146
  Day 43 | 79.9 [79.9 to 79.9] | 5977.3 [5456.5 to 6547.9]
  Day 57: number analyzed (Participants) | 50 | 146
  Day 57 | 79.9 [79.9 to 79.9] | 1734.7 [1582.8 to 1901.2]
  Day 209: number analyzed (Participants) | 12 | 144
  Day 209 | 79.9 [79.9 to 79.9] | 741.3 [630.2 to 872.0]
  Day 394: number analyzed (Participants) | 7 | 129
  Day 394 | 79.9 [79.9 to 79.9] | 248.0 [202.8 to 303.2]

23. Secondary Outcome: GMFR of Serum nAb Against SARS-CoV-2 on Days 29, 43, 57, 209, and 394
Description: The GMFR was calculated as the ratio of the post-vaccination titer level to the baseline titer level. Where baseline was defined as the last measurement taken before the first dose of study intervention. GMFR of serum nAb against SARS-CoV-2 was measured by assay specific to wild-type virus.
Time Frame: At Days 29, 43, 57, 209, and 394
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
fold change
  Day 29: number analyzed (Participants) | 50 | 139
  Day 29 | 1.0 [1.0 to 1.0] | 2.5 [2.1 to 3.0]
  Day 43: number analyzed (Participants) | 50 | 146
  Day 43 | 1.0 [1.0 to 1.0] | 74.8 [68.3 to 82.0]
  Day 57: number analyzed (Participants) | 50 | 146
  Day 57 | 1.0 [1.0 to 1.0] | 21.7 [19.8 to 23.8]
  Day 209: number analyzed (Participants) | 12 | 144
  Day 209 | 1.0 [1.0 to 1.0] | 9.3 [7.9 to 10.9]
  Day 394: number analyzed (Participants) | 7 | 129
  Day 394 | 1.0 [1.0 to 1.0] | 3.1 [2.5 to 3.8]

24. Secondary Outcome: SCR of Serum nAb Against SARS-CoV-2 on Days 29, 43, 57, 209, and 394
Description: SCR was defined at percentage of participants with a change from below the LOD or LLOQ to equal to or above LLOQ, OR, >=4-fold rises from baseline. LLOQ= 159.79 and ULOQ= 11173.11. Baseline was defined as the last measurement taken before the first dose of study intervention. SCR of serum nAb against SARS-CoV-2 was measured by assay specific to wild-type virus.
Time Frame: At Days 29, 43, 57, 209, and 394
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-919 0.5 mL
Number analyzed (Participants) | 50 | 147
percentage of participants
  Day 29: number analyzed (Participants) | 50 | 139
  Day 29 | 0.0 [0.0 to 7.1] | 56.1 [47.5 to 64.5]
  Day 43: number analyzed (Participants) | 50 | 146
  Day 43 | 0.0 [0.0 to 7.1] | 100.0 [97.5 to 100.0]
  Day 57: number analyzed (Participants) | 50 | 146
  Day 57 | 0.0 [0.0 to 7.1] | 100.0 [97.5 to 100.0]
  Day 209: number analyzed (Participants) | 12 | 144
  Day 209 | 0.0 [0.0 to 26.5] | 94.4 [89.3 to 97.6]
  Day 394: number analyzed (Participants) | 7 | 129
  Day 394 | 0.0 [0.0 to 41.0] | 68.2 [59.4 to 76.1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are AEs that started after the first vaccination on Day 1 up to 365 days after the second vaccination on Day 29 (Day 394)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-919 0.5 mL
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/150
Other Adverse Events (participants affected / at risk) | 21/50 | 144/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | TAK-919 0.5 mL (N=150)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | TAK-919 0.5 mL (N=150)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 50
Body temperature increased (Investigations) | 1 | 60
Chills (General disorders) | 1 | 77
Fatigue (General disorders) | 9 | 97
Headache (Nervous system disorders) | 7 | 74
Induration (General disorders) | 0 | 21
Injection site pain (General disorders) | 4 | 138
Injection site pruritus (General disorders) | 0 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 91
Swelling (General disorders) | 0 | 29
Vaccination site erythema (General disorders) | 0 | 28
Vaccination site lymphadenopathy (General disorders) | 4 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT04677660/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04677660/SAP_001.pdf